CLINICAL TRIAL: NCT06783322
Title: The ARCTIC REWIND Extension Study - Long-term Outcomes of Patients with Rheumatoid Arthritis in Remission
Brief Title: Long-term Outcomes of Patients with Rheumatoid Arthritis in Remission
Status: Not yet recruiting | Type: Observational
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other); The Research Council of Norway (Other); Olav Thon Foundation (Unknown)
Responsible Party: Principal Investigator, Nina Sundlisæter, PhD, Diakonhjemmet Hospital
Other Study IDs: DS-00887
Record Dates: First submitted 2024-12-12; First posted 2025-01-20 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: remission; tapering; drug-free remission; long-term outcomes
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, buffy coat, PBMC, RNA storage tubes and full blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this multi-center prospective observational study is to develop knowledge on how to best personalize treatment and follow-up strategies for patients with RA in remission, with the intention to prevent relapse of disease activity and progression of joint damage and at the same time avoid the use of unnecessary treatment and health resources.

The investigators will perform an extensive evaluation of all patients who participated in the ARCTIC REWIND study 10 and 15 years after they achieved sustained remission and received different treatment strategies.

DETAILED DESCRIPTION:
Rheumatoid Arthritis (RA) is a chronic inflammatory disease that affects 0.5 to 1.0% of the population. In case of ineffective treatment, the inflammation can lead to joint destruction and reduced physical function, as well as affecting internal organs. RA is associated with an increased risk of cardiovascular disease and osteoporosis.

The prognosis for RA has improved significantly over the past two decades, with effective treatment strategies and available drugs allowing a significant proportion of patients to achieve the treatment goal of remission (absence of signs of inflammation). RA has thus become a 'controllable' disease, and the large increase in the number of RA patients in remission leaves a need for improved understanding of how to best treat these patients.

A total of 259 RA patients in sustained remission were included in the ARCTIC REWIND trial. They were randomized to either tapering of DMARDs, or to continue stable DMARD medication, and followed for three years. The current study will provide a 10- and 15-year follow-up on the outcome of all these patients.

The results from the project will add knowledge about the long-term consequences of achieving sustained remission, as well as of experiencing a disease activity flare regarding DMARD use, joint damage progression, functional status and work productivity, and the study will provide novel data on cardiovascular health and other comorbidities in this patient group. Further, the patient perspective on flare will be explored. Such information will be valuable for patients and clinicians to improve shared decision on further treatment, and potentially allow more patients to reduce treatments in an evidence-based manner. Results from the study could influence approaches to the management of RA in the future, as selecting patients who can be switched to remote care (reduce the number of visits the patient has to attend physically).

ELIGIBILITY:
Inclusion Criteria:

* Participation in the ARCTIC REWIND trial
* Patients able and willing to give written informed consent and comply with the requirements of the study protocol

Exclusion Criteria:

* Psychiatric or mental disorders, alcohol abuse, other substance abuse, other factors making adherence to the study protocol impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of men and women with established rheumatoid arthritis who have experienced sustained remission and participated in the ARCTIC REWIND trial. All the 259 patients that entered the ARCTIC REWIND trial are eligible to participate in the extension study.
Sampling Method: Non-Probability Sample
Enrollment: 259 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2034-01 (Estimated); Study Completion 2034-01 (Estimated)

PRIMARY OUTCOMES:
Disease activity remission status | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  Remission status will be assessed according to e.g the disease activity score DAS, the Simplified Disease Activity Index (SDAI) and ACR/EULAR Boolean 2.0 remission.
  DAS includes the ritchie articular index, the swollen joint count (based on 44 joints), the ESR and the Patient's Global Assessment of disease activity on a VAS 0-100 mm (PGA). The following cut-points are used:
  High disease activity: DAS > 3.7; Moderate disease activity: 3.7 ≥ DAS>2.4; Low disease activity: 2.4 ≥ DAS ≥ 1.6; In remission: DAS < 1.6
  The SDAI includes tender and swollen joints (of 28), PGA, PhGA and CRP. According to SDAI, the following cut-points are used:
  High disease activity: SDAI> 26.0; Moderate disease activity: 26.0 ≥ SDAI>11.0; Low disease activity: 11.0 ≥ SDAI > 3.3; In remission: SDAI ≤ 3.3
  ACR/EULAR 2.0 remission is defined as the combination of tender joints ≤ 1, swollen joints ≤ 1, CRP ≤ 1 and patient global assessment ≤ 2 (on a scale 0-10).
Disease Modifying Anti-Rheumatic Drug (DMARD)-free remission | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  The prevalence of DMARD-free remission
Radiographic score (van der Heijde modified Sharp score (vdHSS) | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  Radiographs of hands and feet. The van der Heijde-modified Sharp scoring method will be used, which assesses erosions in 16 joints of each hand (range, 0-5 for each joint) and in 6 joints of each foot (range, 0-10 per joint) and joint space narrowing in 15 joints for each hand and in 6 joints for each foot (range, 0-4 per joint).This gives scores for erosions on a scale from 0 to 280 and joint space narrowing on a scale from 0 to168, thus the total van der Heijde-modified Sharp score ranges from 0 to 448, with higher scores indicating greater joint damage.
Radiographic joint damage progression | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  Radiographs of hands and feet. The van der Heijde-modified Sharp scoring method will be used, which assesses erosions in 16 joints of each hand (range, 0-5 for each joint) and in 6 joints of each foot (range, 0-10 per joint) and joint space narrowing in 15 joints for each hand and in 6 joints for each foot (range, 0-4 per joint).This gives scores for erosions on a scale from 0 to 280 and joint space narrowing on a scale from 0 to168, thus the total van der Heijde-modified Sharp score ranges from 0 to 448, with higher scores indicating greater joint damage.
  The images will be compared to the last corresponding images undertaken in the ARCTIC REWIND trial.
  Progression will be calculated as e.g. annual increase in van der Heijde modified Sharp score ≥ 1 unit.
Disease activity composite measures | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  The following composite measures will be included: disease activity score (DAS), DAS based on 28 joint counts (DAS28), the simplified disease activity index (SDAI) and the clinical disease activity index (CDAI). These are based on tender and swollen joint counts, the PGA, acute phase reactants (except from CDAI), and, for SDAI and CDAI also the PhGA.
  DAS: High disease activity: DAS > 3.7; Moderate disease activity: 3.7 ≥ DAS>2.4; Low disease activity: 2.4 ≥ DAS ≥ 1.6; In remission: DAS < 1.6
  DAS28: High disease activity: DAS28 > 5.1; Moderate disease activity: 5.1 ≥ DAS28>3.2; Low disease activity: 3.2 ≥ DAS28 ≥ 2.6; In remission: DAS28 < 2.6
  CDAI: High disease activity: CDAI > 22.0; Moderate disease activity: 22.0 ≥ CDAI>10.0; Low disease activity: 10.0 ≥ CDAI > 2.8; In remission: CDAI ≤ 2.8
  SDAI: High disease activity: SDAI> 26.0;Moderate disease activity: 26.0 ≥ SDAI>11.0; Low disease activity: 11.0 ≥ SDAI; In remission SDAI ≤ 3.3
Patient reported physical function | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  The Patient-Reported Outcomes Measurement Information (PROMIS) HAQ (Health Assessment Questionnaire ) 20-item short form will be used in this study. Each question has five response options, ranging in value from one to five. To find the total raw score, the sum of the values of the response to each question is calculated, giving a range in scores from 20 to 100 if all questions are answered. The total raw score should be translated into a T-score for each participant (either by standardized conversion tables or using item-level calibrations), which rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD worse than average.

SECONDARY OUTCOMES:
Health-related quality of life | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  EuroQol-5 Dimensions three-level (EQ-5D-3L) is a utility instrument for measurement of health-related quality of life. It comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems (labelled 1-3). They have no arithmetic properties and should not be used to derive a summary score. To derive the summary index score an appropriate value set is required, which provides values (weights) for each health state description according to the preferences of the general population of a country/region
Patient global assessment of disease activity | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  0-100 visual analogue scale (VAS), with higher scores Indicating more disease activity
Physician global assessment of disease activity | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  0-100 visual analogue scale (VAS), with higher scores Indicating more disease activity
Ultrasound inflammation | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  Ultrasound joint inflammation will be assessed by use of a validated 0-3 semi-quantitative scoring system for power Doppler and grey scale with an ultrasound atlas as reference. In the total ultrasound score 32 joints will be included: Bilateral metacarpophalangeal (MCP) joint I-V, radiocarpal joint, distal radioulnar joint, intercarpal joint, elbow, knee, talocrural joint and metatarsophalangeal (MTP) joint I-V, yielding a maximum total score of 96. In addition to the 32 joints the following will be scored: Bilateral proximal Interphalangeal (PIP) 2 and 3 joints, extensor carpi ulnaris tendon and tibialis posterior tendon.
Swollen joint count | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  Assessment of 44 joints
Tender joint count | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  Assessment of 44 tender joints
Tender joints | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  Assessed by Ritchie Articular index
Osteoporosis | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  Assessed by Dual-energy X-ray absorptiometry (DEXA)
Medication use | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  Record of disease modifying antirheumatic drugs including corticosteroids
Physical and mental health | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  This will be assessed by The 36-item Short Form Health Survey (SF-36). The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
  The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health or emotional wellbeing
Patient reported impact of disease | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  Assessed by the Rheumatoid Arthritis Impact of Disease (RAID) score which is a patient-derived composite response index for use in clinical trials in RA. It includes seven domains which are scored between 0 and 10. The domains are given the following relative weights: pain (21%), functional disability (16%), fatigue (15%), emotional well-being (12%), sleep (12%), coping (12%) and physical well-being (12%).
  The range of the final RAID value is 0-10 where higher scores indicate worse status.
Work performance and status | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  Work Productivity and Activity Impairment Questionnaire: WPAI:RA. This is a questionnaire that quantifies health-related work productivity loss for those employed. Work time missed (absentism) and reduced on-the-job effectiveness are expressed in percentages. Overall work productivity loss (abstentism and presentism combined) is also expressed in percentages.
Presence of cardiovascular disease and CVD risk | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  assessed by Systematic Coronary Risk Evaluation 2 (SCORE2), carotid intima-media thickness and plaques, and echocardiography
Erythrocyte Sedimentation Rate (ESR) | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  Blood test
C-reactive protein (CRP) | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  Blood test
Patients reported flare | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  The Outcome Measures in Rheumatology (OMERACT) preliminary Rheumatoid Arthritis Flare Questionnaire version 2.1 will be used. The questionnaire includes information about variables deemed to be of relevance by both patients and health care professionals to describe and define RA flare. It assesses severity and duration of flare, self-management strategies related to flare, pain, function, fatigue, stiffness, participation, coping, and patients' self-assessment of joint tenderness and swelling.
  Patients who classifies themselves as flaring rates the severity on a 11-point Numerical Rating Scale (0-10), the higher score the worse.
Registration of comorbidities | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  Questionnaire about comorbidities, including, but not limited to, cardiovascular/cerebrovascular disease, respiratory disease, diabetes mellitus, hypertension requiring treatment, cancer, fibromyalgia, osteoporosis, depression requiring treatment, joint replacements, hip fractures, and abdominal perforations.
Fatigue | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  Fatigue is self-reported with use of a visual analogue scale that ranges from 0 to 100 mm, with higher scores indicating more severe fatigue.
Joint pain | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  joint pain is self-reported with use of a visual analogue scale that ranges from 0 to 100 mm, with higher scores indicating more severe joint pain
Patient's acceptable symptom state | Assessed at the visit 10- and 15-year after the initial inclusion into the ARCTIC REWIND trial
  Patient's acceptable symptom state

CONTACTS AND LOCATIONS:
Locations (10):
- Norway (10):
  - Ålesund Hospital, Ålesund
  - Haukeland University Hospital, Bergen
  - Vestre Viken Hospital, Drammen
  - Sørlandet Hospital, Kristiansand
  - Revmatismesykehuset, Lillehammer
  - Helgelandssykehuset Mo i Rana, Mo i Rana
  - Østfold Hospital, Moss
  - Diakonhjemmet Hospital, Oslo
  - Martina Hansens Hospital, Sandvika
  - University Hospital of North Norway, Tromsø

IPD SHARING:
Plan to Share IPD: Undecided